CLINICAL TRIAL: NCT05040178
Title: A Non-Interventional Post-Authorization Safety Study (PASS) of Carbaglu® for the Treatment of Hyperammonemia Due to Methylmalonic Acidemia (MMA) and Propionic Acidemia (PA) in Adult and Pediatric Patient Populations
Brief Title: An Observational Study of Carbaglu® for the Treatment of MMA and PA in Adults and Pediatrics
Status: Recruiting | Type: Observational
Sponsor: RECORDATI GROUP (Industry)
Collaborators: Target PharmaSolutions, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: CARBAGLU-RRDUS-PASS-0573; NCT05842837 (obsolete NCT alias)
Record Dates: First submitted 2021-06-16; First posted 2021-09-10 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-04

CONDITIONS: Hyperammonemia; Methylmalonic Acidemia; Propionic Acidemia
Keywords: PA & MMA
MeSH Terms: conditions — Hyperammonemia; Methylmalonic acidemia; Propionic Acidemia | interventions — carglumic acid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Male and Female Adult and Pediatric Participants: Patients treated with Carbaglu for the treatment for hyperammonemia due to Methylmalonic Acidemia (MMA) and Propionic Acidemia (PA)
  Interventions: Drug: Carglumic Acid

INTERVENTIONS:
Drug: Carglumic Acid — Current or previous treatment with Carbaglu, the dose of Carbaglu® prescribed will be determined by the investigator for each individual patient.
  Other Names: Carbaglu®

SUMMARY:
To obtain short-term and long-term clinical safety information, in pediatric and adult patients with PA and MMA treated with Carbaglu®.

DETAILED DESCRIPTION:
This study is being conducted to obtain short-term and long-term clinical safety information from adult and pediatric patients treated for hyperammonemia due to Methylmalonic Acidemia (MMA) and Propionic Acidemia (PA). This is an observational/non-interventional study. Patients will be treated per the prescribing information and routine medical practice.

Only available data will be collected as part of the study including developmental outcomes, details of treatment with Carbaglu® and other treatments for hyperammonemia including dietary and protein management, plasma ammonia levels, pregnancy and maternal complications, adverse effects on the developing fetus and neonate, adverse effects on the infant through first year of life.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent/assent form
2. Prescribed and treated with Carbaglu®
3. Have an established diagnosis of PA or MMA defined as follows:

   * Diagnosed with PA by semi quantitative urine organic acid analysis, defined as presence of elevated methylcitric acid and normal methylmalonic acid levels and no evidence of biotin related disorders in the organic acid analysis; OR
   * Diagnosed with MMA by semi quantitative urine organic acid analysis, defined as elevation of methylmalonic acid and no evidence of vitamin B12 dependent disorder on plasma amino acid analysis (vitamin B12 dependency is defined by documented vitamin B12 responsiveness).

AND/OR

* Confirmation by molecular genetic testing

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with PA or MMA of any age and gender, including pregnant women, are eligible for enrollment in the study as long as they meet the eligibility criteria.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2022-06-30 (Actual); Primary Completion 2032-06-30 (Estimated); Study Completion 2032-06-30 (Estimated)

PRIMARY OUTCOMES:
Effects of Carbaglu® on plasma ammonia levels | Patients treated with Carbaglu® will be managed chronically (out-patient) or acutely (hospital in-patient). In both cases, data will be collected for approximately 1 year following discontinuation of Carbaglu treatment.
  Multiple plasma ammonia levels will be collected only during treatment with Carbaglu® according to prescribing information and routine medical practice in terms of visit frequency.
Adverse Event frequency and severity | Patients treated with Carbaglu® will be managed chronically (out-patient) or acutely (hospital in-patient). In both cases, data will be collected for approximately 1 year following discontinuation of Carbaglu treatment.
  Any Carbaglu® related adverse events will be be collected and reported

SECONDARY OUTCOMES:
Fetal Outcomes and Pregnancy Outcomes | Collection of pregnancy information for patients who becomes pregnant while participating in the trial or at time of enrollment. Pregnancy reports and reports involving neonates and infants up to 1 year of age must be reported to RRD Pharmacovigilance.
  Pregnancy risks including maternal complications, adverse effects on the developing fetus and neonate, and adverse effects on the infant (through the first year of life).

CONTACTS AND LOCATIONS:
Overall Officials: William Ludlum, MD, Study Director — Recordati Rare Diseases Inc; Nicholas Ah Mew, MD, Principal Investigator — Children's National Research Institute
Locations (5):
- United States (5):
  - Children's National Hospital, Washington D.C., District of Columbia
  - University of South Florida, Tampa, Florida
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Riley Children's Hospital, Indianapolis, Indiana
  - Icahn School of Medicine at Mt. Sinai, New York, New York

IPD SHARING:
Plan to Share IPD: Undecided